CLINICAL TRIAL: NCT03795532
Title: Ultraslow Full-power SWL Versus Slow SWL in Renal Stones With High Attenuation Value
Brief Title: Ultraslow SWL Versus Slow SWL for Renal Stones With High Attenuation Value
Acronym: ESWL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSheemy, Associate Professor of Urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16224
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Renal Stones
Keywords: renal stones; SWL; High density stones; Ultraslow SWL; Slow SWL; Ramping; Pause
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultraslow shock wave lithotripsy (SWL) (Active Comparator): SWL at ultraslow rate of 30 SW/min. Power ramping at the first 100 SW from 6 to 18 kv followed by safety pause for two minutes then power ramping from 18 to 22kv during the second 100 SW followed by safety pause for another two minutes. The rest of the session at 22kv (full power).
  Interventions: Procedure: SWL
- Slow power-ramping SWL (Active Comparator): SWL at a slow rate of 60 SW/min. Power ramping from 6 - 10 kv during the first 500 SW then from 11 - 14 kv during the second 500 SW then from 15 - 18 kv during the following 500 SW then from 19 - 22 kv during the remaining 1000 - 1500 SW.
  Interventions: Procedure: SWL

INTERVENTIONS:
Procedure: SWL — Shock wave lithotripsy
  Other Names: ESWL

SUMMARY:
Ultraslow full-power SWL versus slow power-ramping SWL in Renal stones with high attenuation value

DETAILED DESCRIPTION:
To evaluate the efficacy of ultraslow rate of SWL versus slow rate, power ramping SWL for renal stones

ELIGIBILITY:
Inclusion Criteria:

* single Renal stone less than or equal to 3 cm (2 cm for lower calyceal stones)
* radio-opaque stone
* high attenuation value (≥ 1000 HU) stone

Exclusion Criteria:

* Abnormal renal anatomy
* renal insufficiency
* solitary kidney
* coagulopathies
* uncontrolled hypertension
* renal artery or aortic aneurysm
* active urinary tract infection
* pregnancy
* severe skeletal malformations (spinal deformity) precluding proper stone localization
* skin to stone distance (SSD) > 11 cm
* BMI > 30 Kgm/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
stone free rate | 3 months following last session of SWL
  Complete clearance of stones in addition to clinically insignificant residual fragments

SECONDARY OUTCOMES:
Complications rate | 3 months following last session of SWL
  Comparison of rate of complications in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Aref Al-Dessoukey, Study Director — Beni-Suef University
Locations (1):
- Beni-Suef Hospitals, Banī Suwayf, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No